CLINICAL TRIAL: NCT00413816
Title: A Multicenter Study of Anemia in the ICU Patient: Determination of the Israeli Trigger and Post ICU Course
Brief Title: The Israeli Trigger for Blood Transfusions in the ICU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Other Study IDs: 004152
Record Dates: First submitted 2006-12-19; First posted 2006-12-20 (Estimated); Last update posted 2006-12-20 (Estimated); Status verified 2006-10

CONDITIONS: Anemia
Keywords: Anemia; Critically ill
MeSH Terms: conditions — Anemia; Critical Illness

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The purpose of the study is to determine the trigger for blood transfusions in Israeli ICU patients and the possible effects of anemia on the post ICU discharge course.

DETAILED DESCRIPTION:
Anemia is a common problem in critically ill patients admitted to intensive care units (ICUs). The etiology is multifactorial and includes sepsis, overt or occult blood loss (including frequent blood sampling), decreased production of endogenous erythropoietin, and immune-associated functional iron deficiency. In the only large randomized trial addressing the issue of transfusion triggers in the perioperative and critical care setting, the Canadian Transfusion Requirements in Critical Care (TRICC) study documented an overall non significant trend toward decreased 30-day mortality (18.7% vs. 23.3%, P = .11) and significant decreases in mortality among patients who were less acutely ill (8.7% vs. 16.1%, P = .03) in the group treated using a transfusion trigger reflected in a hemoglobin level of 7.0 g/dL compared with a more liberal transfusion group that received 54% more red blood cell (RBC) transfusions. This data suggests that many critically ill patients can tolerate hemoglobin levels as low as 7 g/dL and that a "liberal" RBC transfusion strategy may in fact lead to worse clinical outcomes. Evidence-based transfusion guidelines for critically ill and perioperative patients recommend RBC transfusion when the hemoglobin concentration is less than 7 g/L and transfusion avoidance at values greater than 10 g/ L .

The restrictive blood transfusion policy results in many patients being discharged anemic from the ICU. In a recent Scottish study, 87% of ICU survivors were discharged anemic (defined as a hemoglobin level < 13g/dl in males and 11 g/dl in females), while 24% of males and 27.9% of females had a hemoglobin level < 9 g/dl. While studies have shown that a restrictive blood transfusion policy does not adversely affect the 30- or 60-day mortality , there is no information regarding the effect of anemia on immediate and long term morbidity of ICU survivors. This may be important as anemia has been shown to decrease functional status and quality of life, while treating anemia may improve functional status and decrease morbidity. In addition, it is not known how many of these patients receive blood transfusions following ICU discharge.

In Israel, there are no national guidelines for the administration of red blood cells in the ICU and the national "trigger" is unknown.

* Study Rationale The determination of the ICU "trigger" will determine if the ICU is performing according to presently accepted standards. Determining the effect of anemia after ICU discharge may allow for targeted interventions in particular groups of patients which may improve recovery rates.
* This study is a non-intervention, observational, multi- center study.
* All ICU patients over 18 years of age will be included.
* Demographic data will be collected on admission of the patient to the ICU
* Daily hemoglobin levels (routine morning hemoglobin) and the hemoglobin level which triggered the blood transfusion (if different from the morning level) will be recorded and the number and indication for red blood cell transfusions noted.
* Hemoglobin level will be noted on discharge from the ICU.
* Hemoglobin levels, length of hospital stay and occurrence of complications in the post-ICU period will be noted.

ELIGIBILITY:
Inclusion Criteria:

* all patients admitted to ICU

Exclusion Criteria:

* age < 18 years
* > 20% full thickness burns

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2006-10; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Cohen, Principal Investigator — Rabin Medical Center, Campus Beilinson, Petah Tikva , Israel, 49100
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel